CLINICAL TRIAL: NCT04865185
Title: Effect of Topical Lidocaine on Warm and Cold Sensation in Healthy Individuals - a Randomized Crossover Trial
Brief Title: Effect of Topical Lidocaine on Warm and Cold Sensation in Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: TLH21
Record Dates: First submitted 2021-04-15; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-03

CONDITIONS: Neuropathy;Peripheral; Thermal Hypesthesia
Keywords: Paradoxical Heat Sensations; Thermal Grill Illusion; Lidocaine
MeSH Terms: conditions — Neuritis; Hypesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylocaine spray 100mg/ml (Active Comparator): Topical application
  Interventions: Diagnostic Test: Xylocaine spray 100mg/ml
- Ethanol (Placebo Comparator): Topical application
  Interventions: Diagnostic Test: Ethanol

INTERVENTIONS:
Diagnostic Test: Xylocaine spray 100mg/ml — Topical application
  Arms: Xylocaine spray 100mg/ml
Diagnostic Test: Ethanol — Topical application
  Arms: Ethanol

SUMMARY:
The purpose of the present study is to systematically test the occurrence of paradoxical and illusory responses to cold and warm stimuli in healthy volunteers with artificial sensory loss.

DETAILED DESCRIPTION:
Efficient thermal sensation is important for adequate behavioral response to cold or warm stimuli and early signs of neuropathy can be changes in the thermal sensation.

Alterations in thermal perception can results in paradoxical heat sensation (a warm perception when the skin is cooled) or a peculiar/burning sensation when the skin is stiumlated with simultaneous warm and cold (a "thermal grill").

Clarifying the occurrence of these paradoxical and illusory sensations, may help understanding early signs of peripheral neuropathy as well as thermal sensory perception.

The investigators plan to conduct a study on thermal sensory perception using a model of sensory loss in healthy volunteers and systematically test the occurrence of paradoxical heat sensations and responses to the thermal grill.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Age between 18 and 40 years
* Participant is able and willing to give informed consent.

Exclusion Criteria:

* Unable to understand and speak Danish
* Non-cooperative
* Chronic pain or acute pain the past week lasting more than 4 hours or pain on the day of investigation
* Pain medication within the last week
* Medication within the last week that can affect assessment
* Psychiatric or neurological disease and diseases that may affect the assessment
* Sensory disturbances
* History or symptoms of significant diseases (e.g. psychiatric or neurological disease, diseases that may affect the assessment, sensory disturbances, cancer, diabetes mellitus, liver diseases, kidney diseases, cardiovascular diseases)
* Pregnancy or lactation
* Jetlag or sleep deprivation
* Alcohol or drug abuse
* Consumption of cannabis the last 4 weeks and consumption of alcohol in the last 48 hours
* Any abnormality of the skin or of vascular origin at application site
* History of hypersensitivity to lidocaine, other amide-type anesthetics, or other contents of the lidocaine or vehicle

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Paradoxical heat sensation (PHS) | 45 minutes
  Number of PHS responders on arm treated with lidocaine 45 minutes after drug application and Number of PHS responders on arm treated with ethanol 45 minutes after drug application

SECONDARY OUTCOMES:
Thermal Grill (TG) | 75 minutes
  Number of TG responders on arm treated with lidocaine 75 minutes after drug application and Number of TG responders on arm treated with ethanol 75 minutes after drug application
Quality of the Thermal Grill (TG) | 75 minutes
  The participants are asked whether the stimulus is burning, hot, warm, neutral, cold, or freezing cold after the TG-condition (warm and cold), only warm or only cold on arm treated with lidocaine 75 minutes after drug application The participants are asked whether the stimulus is burning, hot, warm, neutral, cold, or freezing cold after the TG-condition (warm and cold) or only warm or only cold on arm treated with ethanol 75 minutes after drug application
Pain intensity of the Thermal Grill (TG) | 90 minutes
  The participants are asked to rate the intensity of pain on a visual analog scale (VAS) 0-100 (0 no pain; 100 worst pain imaginable) after the TG-condition (warm and cold), only warm or only cold on arm treated with lidocaine 90 minutes after drug application The participants are asked to rate the intensity of pain on a VAS 0-100 (0 no pain; 100 worst pain imaginable) after the TG-condition (warm and cold), only warm or only cold on arm treated with ethanol 90 minutes after drug application
Intensity of unpleasantness of the Thermal Grill (TG) | 95 minutes
  The participants are asked to rate the intensity of unpleasantness on a VAS 0-100 (0 no unpleasantness; 100 worst unpleasantness imaginable) after the TG-condition (warm and cold), only warm or only cold on arm treated with lidocaine 95 minutes after drug application The participants are asked to rate the intensity of unpleasantness on a VAS 0-100 (0 no unpleasantness; 100 worst unpleasantness imaginable) after the TG-condition (warm and cold), only warm or only cold on arm treated with ethanol 95 minutes after drug application
Intensity of cold of the Thermal Grill (TG) | 95 minutes
  The participants are asked to rate the intensity of unpleasantness on a VAS 0-100 (0 no cold; 100 extremely cold ) after the TG-condition (warm and cold), only warm or only cold on arm treated with lidocaine 95 minutes after drug application
  The participants are asked to rate the intensity of unpleasantness on a VAS 0-100 (0 no cold; 100 extremely cold ) after the TG-condition (warm and cold), only warm or only cold on arm treated with ethanol 95 minutes after drug application
Intensity of warm of the Thermal Grill (TG) | 95 minutes
  The participants are asked to rate the intensity of unpleasantness on a VAS 0-100 (0 no warm; 100 extremely warm ) after the TG-condition (warm and cold), only warm or only cold on arm treated with lidocaine 95 minutes after drug application
  The participants are asked to rate the intensity of unpleasantness on a VAS 0-100 (0 no warm; 100 extremely warm ) after the TG-condition (warm and cold), only warm or only cold on arm treated with ethanol 95 minutes after drug application
Paradoxical heat sensation (PHS) | 30 minutes before drug application
  Number of PHS responders at baseline without any treatment, 30 minutes before drug application
Thermal Grill (TG) | 20 minutes before drug application
  Number of TG responders at baseline without any treatment 20 minutes before drug application

OTHER OUTCOMES:
Thermal thresholds | 45 minutes
  Detection- and pain thresholds for cold, warm (degrees) stimuli at baseline without any treatment
  Detection- and pain thresholds for cold, warm (degrees) stimuli on arm treated with lidocaine 45 minutes after drug application
  Detection- and pain thresholds for cold, warm (degrees) stimuli on arm treated with ethanol 45 minutes after drug application
Paradoxical heat sensation (PHS) using a modified protocol | 100 minutes
  Number of PHS responders if the skin is heated or cooled prior the test at baseline without any treatment Number of PHS responders if the skin is heated or cooled prior the test on arm treated with lidocaine 100 minutes after drug application Number of PHS responders if the skin is heated or cooled prior the test on arm treated with ethanol 100 minutes after drug application
Mechanical thresholds | 45 minutes
  Detection- and pain thresholds for mechanical (mNewton) stimuli at baseline without any treatment
  Detection- and pain thresholds for mechanical (mNewton) stimuli on arm treated with lidocaine 45 minutes after drug application
  Detection- and pain thresholds for mechanical (mNewton) stimuli on arm treated with ethanol 45 minutes after drug application

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L Schaldemose, MD, Principal Investigator — Danish Pain Research Center, Aarhus University
Locations (1):
- Danish Pain Research Center, Aarhus University, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04865185/SAP_000.pdf